CLINICAL TRIAL: NCT00332293
Title: An Evaluation of the Safety and Efficacy of Moxifloxacin AF Ophthalmic Solution 0.5% for the Treatment of Bacterial Conjunctivitis in India
Brief Title: AL-15469A for the Treatment of Bacterial Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-04-40
Record Dates: First submitted 2006-05-31; First posted 2006-06-01 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2012-03

CONDITIONS: Bacterial Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — Alkalies; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Moxifloxacin (Experimental)
  Interventions: Drug: Moxifloxacin Alternative Formulation Ophthalmic Solution 0.5%
- VIGAMOX (Active Comparator)
  Interventions: Drug: Moxifloxacin hydrochloride ophthalmic solution 0.5% as base

INTERVENTIONS:
Drug: Moxifloxacin Alternative Formulation Ophthalmic Solution 0.5% — 1 drop into the conjunctival sac of both eyes 3 times a day for 3 days
  Arms: Moxifloxacin
Drug: Moxifloxacin hydrochloride ophthalmic solution 0.5% as base — 1 drop into the conjunctival sac of both eyes 3 times a day for 3 days
  Other Names: VIGAMOX
  Arms: VIGAMOX

SUMMARY:
The purpose of the study is to determine whether AL-15469A is safe and effective in the treatment of bacterial conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* signs and symptoms of bacterial conjunctivitis
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* under 1 mo. age
* Other protocol-defined exclusion criteria may apply

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 695 (Actual)
Dates: Start 2006-05; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Clinical cure and microbiological success

SECONDARY OUTCOMES:
Individual signs and symptoms of bacterial conjunctivitis at each visit

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon for Trial Locations, Fort Worth, Texas, United States

REFERENCES:
- [Result] Tauber S, Cupp G, Garber R, Bartell J, Vohra F, Stroman D. Microbiological efficacy of a new ophthalmic formulation of moxifloxacin dosed twice-daily for bacterial conjunctivitis. Adv Ther. 2011 Jul;28(7):566-74. doi: 10.1007/s12325-011-0037-x. Epub 2011 Jun 14. PMID 21681652